CLINICAL TRIAL: NCT01119105
Title: A Phase II, Multi-center, Randomized, Double-blind Study Comparing the Safety and Efficacy of Two Doses of BC-3781 Versus Vancomycin in Patients With Acute Bacterial Skin and Skin Structure Infection
Brief Title: Study Comparing the Safety and Efficacy of Two Doses of BC-3781 vs Vancomycin in Patients With Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAB-BC-3781-2001
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Bacterial Infections; Infection
Keywords: acute bacterial skin and skin structure infection; bacteria
MeSH Terms: conditions — Bacterial Infections; Infections | interventions — lefamulin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BC-3781 dose 100mg (Experimental)
  Interventions: Drug: BC-3781
- BC-3781 dose 150mg (Experimental)
  Interventions: Drug: BC-3781
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: BC-3781 — BC-3781 dose 100mg is administered as i.v. infusion every 12 h for 5 to 14 days depending on the clinical response.
  Arms: BC-3781 dose 100mg
Drug: BC-3781 — BC-3781 dose 150mg is administered as i.v. infusion every 12 h for 5 to 14 days depending on the clinical response.
  Arms: BC-3781 dose 150mg
Drug: Vancomycin — Vancomycin is administered as i.v. infusion every 12 h for 5 to 14 days depending on the clinical response.
  Arms: Vancomycin

SUMMARY:
This is a Phase II, multi-center, randomized, double-blind study comparing the safety and efficacy of two doses of BC-3781 versus vancomycin in patients with acute bacterial skin and skin structure infection.

DETAILED DESCRIPTION:
The purpose of the study is to determine the efficacy of 2 dose regimens of BC-3781 versus the licensed medicinal product vancomycin over 5 to 14 days. The population in this study will be patients with an acute bacterial skin and skin structure infection (ABSSSI) and they will receive treatment with one of two doses of BC-3781 or vancomycin, a standard treatment for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18
* Documented acute bacterial skin and skin structure infection

Exclusion Criteria:

* Uncomplicated skin and skin structure infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2011-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T. Prince, Dr., Study Chair — Nabriva Therapeutics AG
Locations (9):
- United States (9):
  - BC-3781 Study Center 002, Chula Vista, California
  - BC-3781 Study Center 001, La Mesa, California
  - BC-3781 Study Center 003, Oceanside, California
  - BC-3781 Study Center 012, Columbus, Georgia
  - BC-3781 Study Center 018, Savannah, Georgia
  - BC-3781 Study Center 021, Baton Rouge, Louisiana
  - BC-3781 Study Center 023, Lafayette, Louisiana
  - BC-3781 Study Center 004, Butte, Montana
  - BC-3781 Study Center 016, Somers Point, New Jersey

REFERENCES:
- [Derived] Rubino CM, Xue B, Bhavnani SM, Prince WT, Ivezic-Schoenfeld Z, Wicha WW, Ambrose PG. Population pharmacokinetic analyses for BC-3781 using phase 2 data from patients with acute bacterial skin and skin structure infections. Antimicrob Agents Chemother. 2015 Jan;59(1):282-8. doi: 10.1128/AAC.02033-13. Epub 2014 Oct 27. PMID 25348519

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BC-3781 Dose 100mg | BC-3781 Dose 150mg | Vancomycin
Started | 70 | 72 | 68
Completed | 66 | 66 | 60
Not Completed | 4 | 6 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 5
Not completed — Adverse Event | 1 | 0 | 1
Not completed — study drug missed on 2 consecutive days | 1 | 2 | 1
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | BC-3781 Dose 100mg | BC-3781 Dose 150mg | Vancomycin | Total
Number analyzed (Participants) | 70 | 71 | 66 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 66 | 68 | 63 | 197
  >=65 years | 4 | 3 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (13.07) | 42.2 (13.41) | 40.4 (13.70) | 41.4 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 27 | 73
  Male | 48 | 47 | 39 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 14 | 37
  Not Hispanic or Latino | 59 | 59 | 52 | 170
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 0 | 7
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 9 | 13 | 6 | 28
  White | 56 | 51 | 59 | 166
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Diabetic Status [Count of Participants; unit: Participants]
  Diabetic | 14 | 19 | 10 | 43
  Non-diabetic | 56 | 52 | 56 | 164
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 34 | 31 | 32 | 97
  Past Smoker | 7 | 7 | 11 | 25
  Non-Smoker | 29 | 33 | 23 | 85

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical Response of Success was defined as resolution of the subject's clinical signs and symptoms with no additional antimicrobial therapy required.
Time Frame: Test of Cure (TOC), 7 - 14 days post final treatment
Population: Clinically Evaluable Population: A subset of all randomized patients who met additional pre-defined criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | BC-3781 Dose 100mg | BC-3781 Dose 150mg | Vancomycin
Number analyzed (Participants) | 60 | 54 | 51
Participants
  Success | 54 | 48 | 47
  Failure | 6 | 6 | 4

2. Primary Outcome: Clinical Response
Description: as for outcome 1
Time Frame: Test of Cure (TOC), 7 - 14 days post final treatment
Population: Modified Intent-to-Treat Population: A subset of the Intent-to Treat Population who had a documented Gram-positive pathogen from a blood culture or from a culture of the acute bacterial skin and skin structure infection at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | BC-3781 Dose 100mg | BC-3781 Dose 150mg | Vancomycin
Number analyzed (Participants) | 50 | 51 | 51
Participants
  Success | 41 | 42 | 42
  Failure | 8 | 6 | 6
  Missing | 1 | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from the time of consent through 30 days following the last dose of study medication; approximately 35 to 44 days per participant.
Description: Adverse events were reported for the ITT population (i.e. all patients who received at least one dose of study medication). Treatment-emergent adverse events, defined as adverse events that started on or after the first dose of study medication, are reported. Adverse events were recorded whether or not they were considered to be study drug related.
Arm/Group | BC-3781 Dose 100mg | BC-3781 Dose 150mg | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/70 | 2/71 | 2/66
Other Adverse Events (participants affected / at risk) | 50/70 | 48/71 | 49/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BC-3781 Dose 100mg (N=70) | BC-3781 Dose 150mg (N=71) | Vancomycin (N=66)
Abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BC-3781 Dose 100mg (N=70) | BC-3781 Dose 150mg (N=71) | Vancomycin (N=66)
Constipation (Gastrointestinal disorders) | 2 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 4
Nausea (Gastrointestinal disorders) | 7 | 7 | 11
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3
Infusion Site Phlebitis (General disorders) | 4 | 2 | 0
Pyrexia (General disorders) | 2 | 3 | 4
Cellulitis (Infections and infestations) | 3 | 4 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 2 | 3
Blood Creatine Phosphokinase Increased (Investigations) | 3 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 3
Headache (Nervous system disorders) | 8 | 13 | 15
Insomnia (Psychiatric disorders) | 1 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 9
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data from the study is confidential information. Sponsor has the right to publish first. Thereafter, PI may publish data from the study, but PI must submit the publication to Sponsor for review at least 60 days prior to publication. Sponsor may remove any confidential and/or proprietary information. If Sponsor's publication is not submitted within 12 months after the study, or if Sponsor decides not to publish, PI may publish the data, subject to Sponsor's rights in the agreement.